CLINICAL TRIAL: NCT07405398
Title: A Study to Train a Machine Learning Algorithm for an Evaluation of the Use of Biometric Data Captured at the Wrist for the Identification of Acute Opioid Use Events and the Quantification of Opioid Withdrawal in Opioid Dependent Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OpiAID (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OA-SBIR-25-01; 4R44DA058474-02 (NIH)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Treatment for Opioid Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm 14 day monitoring period (Experimental): The goal of this real-world, multi-center, outpatient study is to train a machine learning model/algorithm utilizing patient-specific physiological parameters from the OpiAID Strength Band Platform™ can accurately detect MOUD events during the induction phase with a predefined classification success when comparing the True Positive Rate against the False Positive Rate as plotted on a Receiver Operator Curve. In addition to MOUD detection, machine learning will be used to quantify participant withdrawal level from physiological parameters. To demonstrate that withdrawal quantification performs as well or better than current measures used for this purpose the correlation between quantified withdrawal and time since last opioid dose (TSLD) will be computed and compared against the association between SOWS and TSLD in a non-inferiority analysis.
  Prescribing physician must determine appropriate starting dose (titration expected over 2-6 weeks)
  Interventions: Device: Train and evaluate the accuracy and reliability of the Strength Band Platform in identifying acute opioid dosing events from time-stamped biometric data collected from wrist-worn devices.

INTERVENTIONS:
Device: Train and evaluate the accuracy and reliability of the Strength Band Platform in identifying acute opioid dosing events from time-stamped biometric data collected from wrist-worn devices. — Subjects will be fitted with the wearable device (Samsung Galaxy Watch) for the purpose of data communication and will be instructed to wear the device continuously, except when charging the watch, showering or any activity in which submersion in water is required. Participants will wear the device for 14 days.
  Study subjects will be responsible for:
  * Wearing the Samsung Galaxy watch daily except when charging the watch, showering or any activity in which submersion in water is required
  * Charging the Samsung Galaxy watch daily
  * Answering prompts on the Samsung Galaxy watch
  * Answering the daily SOWS questionnaire(s)

SUMMARY:
To train a machine learning model/algorithm for an evaluation of the use of biometric data captured at the wrist for the identification of acute opioid use events and the quantification of opioid withdrawal in opioid dependent individuals.

DETAILED DESCRIPTION:
The goal of this real-world, multi-center, outpatient study is to train a machine learning model/algorithm utilizing patient-specific physiological parameters from the OpiAID Strength Band Platform™ can accurately detect MOUD events during the induction phase with an 80% classification success when comparing the True Positive Rate against the False Positive Rate as plotted on a Receiver Operator Curve. In addition to MOUD detection, machine learning will be used to quantify participant withdrawal level from physiological parameters. To demonstrate that withdrawal quantification performs as well or better than current measures used for this purpose the correlation between quantified withdrawal and time since last opioid dose (TSLD) will be computed and compared against the association between SOWS and TSLD in a non-inferiority analysis.

ELIGIBILITY:
Inclusion Criteria:

Male or female Age ≥22 years at signing of informed consent Patients with a DSM-5 diagnosis of OUD who are eligible for MOUD induction with methadone or buprenorphine

Exclusion Criteria:

Sleeve tattoo covering the wrist Subject unable to independently navigate and operate smartwatch applications Subject not proficient with written and spoken English Subject determined likely to be non-compliant by physician/HCP Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge.

History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.

Subject has diminished decision making capability

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Classification | 14 days
  Accurate algorithm-based classification of acute opioid dosing events in patients receiving treatment for opioid use disorder.

CONTACTS AND LOCATIONS:
Overall Officials: David MacQueen, PhD, Study Chair — OpiAID
Locations (3):
- United States (3):
  - Coastal Horizon, Wilmington, North Carolina
  - Community Medical Services, Austin, Texas
  - Community Medical Services, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: Undecided